CLINICAL TRIAL: NCT03262571
Title: Usefulness of Lung Ultrasound in Ambulatory Management of Patients With Chronic Heart Failure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Because at the interim analysis the pre-specified stopping boundary for an overwhelming benefit had been crossed.
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Agricola Eustachio, MD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-LINES
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Chronic Heart Failure; Lung; Congestive; Acute Decompensated Heart Failure
Keywords: Heart failure; Lung ultrasound; B-lines
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A includes patients undergoing lung ultrasound and physical examination.
  Interventions: Diagnostic Test: Lung ultrasound
- Group B (Placebo Comparator): Group B includes patients undergoing physical examination only.
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Duretic therapy is then optimized according to the presence and severity of B-lines in group A.

SUMMARY:
Purpose. The aim of this study is to evaluate whether lung ultrasound, in addition to physical examination, leads to a reduction of the admission rate for acute decompensated heart failure of patients with chronic heart failure (HF) followed in the outpatients heart failure clinic.

Methods. This is a prospective randomized study. The planned sample size consists of 440 patients with chronic HF.

The inclusion criteria are: (1) male and female aged between 18 and 90 years (2) signed written informed consent (3) history of HF for at least six months, (4) left ventricular ejection fraction < 45%, (5) adequate medical therapy for HF for at least two months.

The exclusion criteria are: (1) concomitant enrollment in other clinical studies, or treatment with experimental drugs or devices within 30 days of clinical assessment, (2) inability to undergo to the planned follow-up and procedures (3) documented pulmonary infections (3) interstitial lung disease and class 4 chronic obstructive pulmonary disease according to GOLD classification.

Patients are randomized in two groups: group A, patients undergoing to lung ultrasound and physical examination; and group B, patients undergoing to physical examination only. Patients are evaluated at baseline and after three months with medical history, Quality of Life test, physical examination, blood sample for hematochemical (creatinine, electrolytes, BNP/NTpro-BNP).

The diuretic therapy is then optimized according to the presence and severity of B-lines in group A and physical examination in group B.

Only patients enrolled in group A undergo to a lung ultrasound examination to assess the extent of pulmonary congestion, through its evidence of B-lines. B-lines originate from the contrast between air-filled structures and water-thickened pulmonary interlobular septa. This leads to linear echogenic vertical artefacts that spread from the pleural layers downwards in the screen. The ultrasound examination is performed with a handheld echocardiography device. The physician carries out a scan of the pulmonary fields, from basal towards mid and apical fields, through the midaxillary line while the patient lies supine. The quantification of B-lines is performed according to their extent over the lung fields. All the information are recorded in dedicated forms.

The results are evaluated according to the following criteria. The primary end-point is a significant reduction of hospitalizations for acute decompensated HF in group A during the follow-up period. The secondary end-points are changes of NT-proBNP values, quality of life test (QLT) score and cardiac mortality.

ELIGIBILITY:
Inclusion Criteria:

(1) male and female aged between 18 and 90 years (2) signed written informed consent (3) history of HF for at least six months, (4) left ventricular ejection fraction < 45%, (5) adequate medical therapy for HF for at least two months.

Exclusion Criteria:

(1) concomitant enrollment in other clinical studies, or treatment with experimental drugs or devices within 30 days of clinical assessment, (2) inability to undergo to the planned follow-up and procedures (3) documented pulmonary infections (4) interstitial lung disease, class 4 chronic obstructive pulmonary disease according to GOLD guidelines (5) chronic dialysis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Reduction of hospitalizations for acute decompensated heart failure | 90 days
  Significant reduction of hospitalizations for acute decompensated heart failure in group A during the 90-day follow-up period.

SECONDARY OUTCOMES:
Natriuretic peptides values | 90 days
  Significant reduction of natriuretic peptides values in group A during the 90-day follow-up period.
Quality of life test (QLT) score | 90 days
  Significant reduction of QTL score in group A during the 90-day follow-up period.
Cardiac mortality | 90 days
  Significant reduction of cardiac mortality rate in group A versus group B.

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No